CLINICAL TRIAL: NCT04004936
Title: Reducing Potentially Inappropriate Medication Prescribing for Older Patients: Enhancing Quality of Provider Practices for Older Adults in the Emergency Department (EQUIPPED)
Brief Title: Reducing Potentially Inappropriate Medication Prescribing for Older Patients in the ED
Acronym: EQUIPPED
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: Durham VA Health Care System (U.S. Federal Agency); VA Salt Lake City Health Care System (U.S. Federal Agency); Birmingham, Alabama VA Medical Center (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: IIR 17-236; IIR HX00257-01A1 (Other Grant/Funding Number: VA Health Services Research & Development)
Record Dates: First submitted 2019-06-28; First posted 2019-07-02 (Actual); Results first posted 2024-08-06 (Actual); Last update posted 2024-08-06 (Actual); Status verified 2024-08

CONDITIONS: Aging
Keywords: Emergency Department; Potentially Inappropriate Medications; Inappropriate Prescribing; Quality Improvement; Veteran Health; Older Adults
MeSH Terms: conditions — Emergencies

STUDY DESIGN:
Intervention Model Description: In order to inform a Veterans Affairs (VA) system-wide approach to improve prescribing safety for older Veterans, the investigators will conduct a randomized study to determine best practices for influencing provider prescribing behavior in order to decrease PIMs prescribed for older Veterans at the time of ED discharge. The overall goal of this project is to determine which EQUIPPED implementation strategy (active or passive feedback) is most effective to reduce prescribing of PIMs for older Veterans discharged from the ED. Eight sites will be randomized to either active feedback with individual, in-person academic detailing or passive feedback delivered via an individualized electronic dashboard.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Active Feedback (Active Comparator): EQUIPPED with active provider feedback, implementing one-to-one (1:1) in-person academic detailing from a professional colleague that includes in-person audit, feedback, and peer benchmarking and provide on-site expertise.
  Interventions: Other: EQUIPPED with Active Feedback
- Passive Feedback (Active Comparator): EQUIPPED with passive provider feedback, implementing monthly provider feedback via an electronic dashboard with audit, feedback and peer benchmarking.
  Interventions: Other: EQUIPPED with Passive Feedback

INTERVENTIONS:
Other: EQUIPPED with Active Feedback — Enhancing Quality of Prescribing Practices for Older Adults Discharged from the Emergency Department (EQUIPPED is a multi-component program to reduce the prescribing of potentially inappropriate medications (PIMs) to older adults upon discharge from the Emergency Department (ED). It has three core components: 1) provider education, 2) Electronic Health Record (EHR)-based clinical decision support (CDS) including pharmacy quick order sets to facilitate provider order entry, and 3) provider audit and feedback with peer benchmarking. The active feedback group will receive one-to-one (1:1) in-person academic detailing from a professional colleague that includes in-person audit, feedback, and peer benchmarking and provide on-site expertise.
  Arms: Active Feedback
Other: EQUIPPED with Passive Feedback — Enhancing Quality of Prescribing Practices for Older Adults Discharged from the Emergency Department (EQUIPPED is a multi-component program to reduce the prescribing of potentially inappropriate medications (PIMs) to older adults upon discharge from the Emergency Department (ED). It has three core components: 1) provider education, 2) Electronic Health Record (EHR)-based clinical decision support (CDS) including pharmacy quick order sets to facilitate provider order entry, and 3) provider audit and feedback with peer benchmarking. The passive feedback group will receive monthly provider feedback via an electronic dashboard with audit, feedback and peer benchmarking.
  Arms: Passive Feedback

SUMMARY:
This research is being conducted to learn which implementation strategy of EQUIPPED is most effective to improve prescribing practices of ED providers toward older Veterans and determine the factors influencing implementation of this program to reduce the prescribing of PIMs to older adults upon discharge from the ED. The study has three research aims. The procedures for these research aims are described below:

* Aim 1 - Examining the Impact of Passive Provider Feedback vs. Active Provider Feedback Through a Randomized Trial
* Aim 2 - Determination of Factors Affecting Organizational Adoption of EQUIPPED
* Aim 3 - Micro-Costing the Active and Passive Feedback Versions of the EQUIPPED Intervention

DETAILED DESCRIPTION:
Enhancing Quality of Prescribing Practices for Older Adults Discharged from the Emergency Department (EQUIPPED is a multi-component program to reduce the prescribing of potentially inappropriate medications (PIMs) to older adults upon discharge from the Emergency Department (ED). It has three core components: 1) provider education, 2) Electronic Health Record (EHR)-based clinical decision support (CDS) including pharmacy quick order sets to facilitate provider order entry, and 3) provider audit and feedback with peer benchmarking. In order to inform a Veterans Affairs (VA) system-wide approach to improve prescribing safety for older Veterans, the investigators will conduct a study to determine best practices for influencing provider prescribing behavior in order to decrease PIMs prescribed for older Veterans at the time of ED discharge. The overall goal of this project is to determine which EQUIPPED implementation strategy (active or passive feedback) is most effective to reduce prescribing of PIMs for older Veterans discharged from the ED.

ELIGIBILITY:
Inclusion Criteria:

* Prescribers at VA Medical Centers that are implementing EQUIPPED
* Members of the EQUIPPED implementation team at enrolled sites

Exclusion Criteria:

* Providers at VA Medical Centers that are not part of the upcoming EQUIPPED implementation trial.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2024-12-31 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Camille Vaughan, MD MS, Principal Investigator — Atlanta VA Medical and Rehab Center, Decatur, GA; George Lee Jackson, PhD MHA, Principal Investigator — Durham VA Medical Center, Durham, NC
Locations (4):
- United States (4):
  - Birmingham VA Medical Center, Birmingham, AL, Birmingham, Alabama
  - Atlanta VA Medical and Rehab Center, Decatur, GA, Decatur, Georgia
  - Durham VA Medical Center, Durham, NC, Durham, North Carolina
  - VA Salt Lake City Health Care System, Salt Lake City, UT, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No
A de-identified, anonymized dataset will be created and shared.

REFERENCES:
- [Result] Burningham Z, Chen W, Sauer BC, Richter Lagha R, Hansen J, Huynh T, Patel S, Leng J, Halwani A, Kramer BJ. VA Geriatric Scholars Program's impact on prescribing potentially inappropriate medications. Am J Manag Care. 2019 Sep;25(9):425-430. PMID 31518091
- [Result] Peters CB, Hansen JL, Halwani A, Cho ME, Leng J, Huynh T, Burningham Z, Caloyeras J, Matsuda T, Sauer BC. Validation of Algorithms Used to Identify Red Blood Cell Transfusion Related Admissions in Veteran Patients with End Stage Renal Disease. EGEMS (Wash DC). 2019 Jul 3;7(1):23. doi: 10.5334/egems.257. PMID 31304183
- [Result] Burningham Z, Jackson GL, Kelleher J, Stevens M, Morris I, Cohen J, Maloney G, Vaughan CP. The Enhancing Quality of Prescribing Practices for Older Veterans Discharged From the Emergency Department (EQUIPPED) Potentially Inappropriate Medication Dashboard: A Suitable Alternative to the In-person Academic Detailing and Standardized Feedback Reports of Traditional EQUIPPED? Clin Ther. 2020 Apr;42(4):573-582. doi: 10.1016/j.clinthera.2020.02.013. Epub 2020 Mar 25. PMID 32222360
- [Result] Lewinski AA, Crowley MJ, Miller C, Bosworth HB, Jackson GL, Steinhauser K, White-Clark C, McCant F, Zullig LL. Applied Rapid Qualitative Analysis to Develop a Contextually Appropriate Intervention and Increase the Likelihood of Uptake. Med Care. 2021 Jun 1;59(Suppl 3):S242-S251. doi: 10.1097/MLR.0000000000001553. PMID 33976073
- [Result] Chien HC, Morreall D, Patil V, Rasmussen KM, Yong C, Li C, Passey DG, Burningham Z, Sauer BC, Halwani AS. Treatment Patterns and Outcomes in a Nationwide Cohort of Older and Younger Veterans with Waldenstrom Macroglobulinemia, 2006-2019. Cancers (Basel). 2021 Apr 4;13(7):1708. doi: 10.3390/cancers13071708. PMID 33916545
- [Result] Passey D, Healy R, Qualls J, Hamilton CJ, Tilley E, Burningham Z, Sauer B, Halwani A. Development and implementation of a pharmacist-led telehealth medication management program for veterans receiving oral antineoplastic therapies through the MISSION Act. Am J Health Syst Pharm. 2022 May 24;79(11):835-843. doi: 10.1093/ajhp/zxac023. PMID 35084462
- [Result] Friedman DR, Patil V, Li C, Rassmussen KM, Burningham Z, Hamilton-Hill S, Kelley MJ, Halwani AS. Integration of Patient-Reported Outcome Measures in the Electronic Health Record: The Veterans Affairs Experience. JCO Clin Cancer Inform. 2022 Feb;6:e2100086. doi: 10.1200/CCI.21.00086. PMID 35290072
- [Result] Burningham Z, Jackson GL, Kelleher JL, Morris I, Stevens MB, Cohen J, Maloney G, Sauer BC, Halwani AS, Chen W, Vaughan CP. Use of a Medication Safety Audit and Feedback Tool in the Emergency Department Is Affected by Prescribing Characteristics. Appl Clin Inform. 2023 Aug;14(4):684-692. doi: 10.1055/s-0043-1771393. Epub 2023 Aug 30. PMID 37648222

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Active Feedback | Passive Feedback
Started | 36 | 38
Completed | 36 | 38
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Participants were EQUIPPED implementation team members or providers at EQUIPPED implementation sites.
Groups:
- Total: Total of all reporting groups
Arm/Group | Active Feedback | Passive Feedback | Total
Number analyzed (Participants) | 36 | 38 | 74
Age, Categorical [Count of Participants; unit: Participants] — Population: Age was self-reported and not reported by all participants
  Participants
    number analyzed (Participants) | 28 | 30 | 58
    <=18 years | 0 | 0 | 0
    Between 18 and 65 years | 24 | 30 | 54
    >=65 years | 4 | 0 | 4
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Self-reported gender, not required to report
  Participants
    number analyzed (Participants) | 27 | 32 | 59
    Female | 12 | 22 | 34
    Male | 15 | 10 | 25
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 21 | 25 | 46
  Unknown or Not Reported | 14 | 13 | 27
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 2 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 18 | 21 | 39
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 15 | 14 | 29
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 36 | 38 | 74

OUTCOME MEASURES:

1. Primary Outcome: Percentage of PIMs Prescribed
Description: Percentage of prescriptions that are PIMS (potentially inappropriate medications) as defined according to the Beers criteria prescribed to adults aged 65 and older and discharged from the ED.
Time Frame: 12-Months Post Implementation of EQUIPPED
Population: Discharge prescriptions for Veterans 65 and older at EQUIPPED implementation sites
Measure: Count of Units; unit: Prescriptions
Units Other Than Participants: Prescriptions
Arm/Group | Active Feedback | Passive Feedback
Number analyzed (Participants) | 36 | 38
Number analyzed (Prescriptions) | 23648 | 36795
Prescriptions | 1,672 | 2,979

2. Secondary Outcome: Impact of EQUIPPED on Behavior Change and Factors Impacting Implementation
Description: Prescribers at participating EDs will be asked to complete a brief survey at baseline, 6, and 12 months to assess key components of the social cognitive factors that we expect to be impacted by the intervention. Interviews will be conducted with EQUIPPED implementation team members to assess implementation facilitators and barriers.
Time Frame: 12-Months After the Delivery of the First EQUIPPED Report
Reporting Status: Not Posted, anticipated posting 2024-12

3. Secondary Outcome: Micro-Costing the Active and Passive Feedback Versions of the EQUIPPED Intervention
Description: Micro-costing of the intervention will be done to learn details of specific factors that may impact the cost of the intervention to the organization.
Time Frame: 12-Months Post Implementation of EQUIPPED
Reporting Status: Not Posted, anticipated posting 2024-12

ADVERSE EVENTS:
Time Frame: AEs, SAEs, and UAPs were collected from the time at study entry until the end of study participation (an average of 1 years, 6 months).
Description: Adverse events were related to distress from survey questions or data breaches.
Arm/Group | Active Feedback | Passive Feedback
All-Cause Mortality (participants affected / at risk) | 0/36 | 0/38
Serious Adverse Events (participants affected / at risk) | 0/36 | 0/38
Other Adverse Events (participants affected / at risk) | 0/36 | 0/38

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2021-06-25): https://cdn.clinicaltrials.gov/large-docs/36/NCT04004936/Prot_000.pdf
  • Statistical Analysis Plan (2018-08-28): https://cdn.clinicaltrials.gov/large-docs/36/NCT04004936/SAP_001.pdf